CLINICAL TRIAL: NCT01733368
Title: Observational Study to Evaluate the Management of Patients Resynchronized With the QuartetTM LV Quadripolar Lead
Brief Title: QUARTO-II Study to Evaluate the Management of Patients Resynchronized With the QuartetTM LV Quadripolar Lead
Acronym: QUARTO-II
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: CR-1 2-015-SP-HF
Record Dates: First submitted 2012-10-02; First posted 2012-11-27 (Estimated); Results first posted 2018-03-01 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Heart Failure
Keywords: CRT; Optimization; Responders
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Optimization and evolution of the patient will be evaluated over 6 months after the implant.

DETAILED DESCRIPTION:
Patient will be enrolled into the study after Informed Consent signature and CRT-D+quadripolar (QuartetTM) LV lead.

ELIGIBILITY:
Inclusion Criteria:

* Patient with implanted CRT-D device and a QuartetTM quadripolar lead by St. Jude Medical in the left ventricle.
* Patient with an echocardiographic study performed during 1 month prior to the implant and in whom End Systolic Volume of the Left Ventricle (LVESV) has been measured
* Patients who have granted their informed consent.
* Patients above 18 years.

Exclusion Criteria:

* Patients that have been previously resynchronized.
* Patients with aortic stenosis or aortic valve prosthesis
* Patients who are or may potentially be pregnant.
* Patients with a life expectancy <12 months.
* Patients who cannot attend the monitoring visits established by the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heart failure patients
Sampling Method: Non-Probability Sample
Enrollment: 198 (Actual)
Dates: Start 2012-11; Primary Completion 2015-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Javier Alzueta, MD, Principal Investigator — Hospital Clínico Universitario Virgen de la Victoria
Locations (1):
- Hospital Universitario Virgen de la Victoria, Málaga, Spain

IPD SHARING:
Plan to Share IPD: No
No plan

RESULTS

PARTICIPANT FLOW:
Groups:
- Quadripolar Left Ventricular Lead (Quartet Lead): Patients implanted with a Cardiac Resynchronization Therapy Defibrillator (CRT-D) device and the Quartet Left Ventricular (LV) quadripolar lead
Period: Overall Study
Arm/Group | Quadripolar Left Ventricular Lead (Quartet Lead)
Started | 198
Completed | 167
Not Completed | 31

BASELINE CHARACTERISTICS:
Arm/Group | Quadripolar Left Ventricular Lead (Quartet Lead)
Number analyzed (Participants) | 198
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.01 (10.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52
  Male | 146
New York Heart Association (NYHA) Classification [Count of Participants; unit: Participants] — The NYHA Functional Classification provides a simple way of classifying the extent of heart failure:
  I Cardiac disease, but no symptoms and no limitation in ordinary physical activity.
  II Mild symptoms and slight limitation during ordinary activity. III Marked limitation in activity due to symptoms, even during less-than-ordinary activity. Comfortable only at rest.
  IV Severe limitations. Experiences symptoms even while at rest.
  Participants
    NYHA I | 5
    NYHA II | 77
    NYHA III | 111
    NYHA IV | 5
Cardiovascular Etiology: Ischemic, Non-ischemic [Count of Participants; unit: Participants]
  Ischemic | 80
  Non-ischemic | 118
QRS Duration [Mean (Standard Deviation); unit: miliseconds (ms)] | 168 (22.22)
QRS Morphology [Count of Participants; unit: Participants]
  Left Bundle Branch Block (LBBB) | 168
  Right Bundle Branch Block (RBBB) | 20
  Interventricular Conduction Delay (IVCD) | 8
  Unknown | 2
Ejection Fraction (EF) [Mean (Standard Deviation); unit: percentage (%)] | 26.87 (7.38)
Left Ventricular End Systolic Volume (LVESV) [Mean (Standard Deviation); unit: milliliters (ml)] | 155.17 (75.10)

OUTCOME MEASURES:

1. Primary Outcome: Number of Responder Patients (Structural Remodelling)
Description: Structural remodelling is defined as a reduction >15% in Left Ventricle End Systolic Volume (LVESV), measured 6 months after implant.
Time Frame: 6 months after implant
Population: Patients with the 6-month follow-up completed and echocardiographic measurements available
Measure: Count of Participants; unit: Participants
Arm/Group | Quadripolar Left Ventricular Lead (Quartet Lead)
Number analyzed (Participants) | 146
Participants | 94

2. Primary Outcome: Safety Outcomes in CRT Responders and Non-Responders
Description: * Mortality rate,
  * Rate of cardiovascular hospitalizations and for any cause or
  * Combined endpoint (death and all-cause hospitalization)
Time Frame: 6 months after implant
Population: Patients experiencing clinical safety event prior to the 6-month follow-up visit.
Measure: Count of Participants; unit: Participants
Groups:
- 6-Month CRT Responder: Patients implanted with a Cardiac Resynchronization Therapy Defibrillator (CRT-D) device and the Quartet Left Ventricular (LV) quadripolar lead and classified as a responder at 6 months of follow-up.
- 6-Month CRT Non-Responder: Patients implanted with a Cardiac Resynchronization Therapy Defibrillator (CRT-D) device and the Quartet Left Ventricular (LV) quadripolar lead and classified as a non-responder at 6 months of follow-up.
Arm/Group | 6-Month CRT Responder | 6-Month CRT Non-Responder
Number analyzed (Participants) | 94 | 58
Participants
  Death | 0 | 6
  All-cause hospitalization | 17 | 16
  Deaths & Hospitalizations | 17 | 20

3. Secondary Outcome: Number of Responder Patients With Non-conventional Left Ventricular Pacing Vector
Description: Response is defined as a reduction >15% in LVESV, measured 6 months after implant.
  Non-conventional pacing vectors are the pacing vectors exclusive to the Quartet LV quadripolar lead, not available in the conventional bipolar leads.
Time Frame: 6 months after implant
Population: Patients with the 6-month follow-up completed, echocardiographic measurements available and programmed with non-conventional LV pacing vector
Measure: Count of Participants; unit: Participants
Arm/Group | Quadripolar Left Ventricular Lead (Quartet Lead)
Number analyzed (Participants) | 59
Participants | 38

4. Secondary Outcome: Number of Responder Patients With Conventional Left Ventricular Pacing Vector
Description: Response is defined as a reduction >15% in LVESV, measured 6 months after implant.
  Conventional pacing vectors are the pacing vectors available both in the Quartet LV quadripolar lead and in the conventional bipolar leads.
Time Frame: 6 months after implant
Population: Patients with the 6-month follow-up completed, echocardiographic measurements available and programmed with a conventional pacing vector
Measure: Count of Participants; unit: Participants
Arm/Group | Quadripolar Left Ventricular Lead (Quartet Lead)
Number analyzed (Participants) | 87
Participants | 56

ADVERSE EVENTS:
Time Frame: 6 months after CRT implant
Arm/Group | Quadripolar Left Ventricular Lead (Quartet Lead)
All-Cause Mortality (participants affected / at risk) | 6/198
Serious Adverse Events (participants affected / at risk) | 50/198
Other Adverse Events (participants affected / at risk) | 15/198
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Quadripolar Left Ventricular Lead (Quartet Lead) (N=198)
Acute Calculous Cholecystitis (Hepatobiliary disorders) | 1
Atrial or Ventricular arrhythmia (Cardiac disorders) | 11
Bleeding/Hematoma (Surgical and medical procedures) | 3
Cardiac arrest and death (Cardiac disorders) | 1
Cardiac Tamponade (Cardiac disorders) | 1
Death (Cardiac disorders) | 2
Diverticulitis (Gastrointestinal disorders) | 1
Exacerbacion of Heart Failulre (Cardiac disorders) | 8
Exacerbacion of Heart Failulre and Death (Cardiac disorders) | 1
Malignant tumor (General disorders) | 1
Musculoskeletal non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 1
Myocardial infartion (Cardiac disorders) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2
Rhabdomyolysis due to amiodarone and statins treatment (Musculoskeletal and connective tissue disorders) | 1
stroke (Cardiac disorders) | 1
Cardiac perforation (Surgical and medical procedures) | 1
Elevated Pacing Thresholds (Product Issues) | 1
Infection (Surgical and medical procedures) | 2
Lead Dislodgement (Product Issues) | 10
Phrenic Nerve/Diaphragmatic/Extracardiac stimulation (Product Issues) | 1
Sepsis and Death (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Quadripolar Left Ventricular Lead (Quartet Lead) (N=198)
Upgrade of the device to DDD by adding atrial lead (Surgical and medical procedures) | 1
Shiver and physical discomfort during implant (Surgical and medical procedures) | 1
Bleeding/Hematoma (Surgical and medical procedures) | 7
carbon dioxide narcosis (Surgical and medical procedures) | 1
Coronary sinus dissection (Surgical and medical procedures) | 1
Inappropriate ATP (Product Issues) | 1
Nause and vomiting (Surgical and medical procedures) | 1
Pain in the implant site (Surgical and medical procedures) | 1
phrenic nerve/diaphragmatic/extracardiac stimulation (Product Issues) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No